CLINICAL TRIAL: NCT02955966
Title: PET/CT Guided Antifungal Stewardship in Invasive Pulmonary Aspergillosis
Acronym: OPTIFIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut Pasteur, Paris France (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P150916; 2016-A00408-43 (Registry Identifier: IDRCB)
Record Dates: First submitted 2016-11-03; First posted 2016-11-04 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Aspergillosis and Haematological Malignancy
Keywords: Aspergillosis; Haematological malignancy; 18F-FDG PET/CT; Biomarkers
MeSH Terms: conditions — Aspergillosis; Hematologic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with invasive pulmonary aspergillosis (Experimental): Blood collection and imaging 18F-FDG-PET/CT
  Interventions: Device: imaging 18F-FDG-PET/CT; Biological: Blood collection

INTERVENTIONS:
Device: imaging 18F-FDG-PET/CT — 18F-FDG PET Scan at Day 0, W6 and W12
Biological: Blood collection — Blood collection at D0, D3, W1, W2, W4, W6, W12, end of treatment.

SUMMARY:
OPTIFIL is a pilot prospective multicenter study based over the hypothesis that the normalization of the functional imaging 18F-FDG-PET/CT during the Invasive pulmonary aspergillosis (IPA) could occur earlier than that of conventional imaging.

This study evaluates the therapeutic response through a systematic 18F-FDG-PET/CT at week 6. The latter response will be correlated with the kinetics of selected biomarkers including antigens (galactomannan, β-D glucans), circulating Aspergillus DNA and anti-Aspergillus host response markers in addition to the conventional imaging tools obtained at weeks 6 and 12.

DETAILED DESCRIPTION:
Invasive pulmonary aspergillosis (IPA) is the 3rd most frequent invasive mycosis in France with a rising incidence and 40% mortality (Bitar, 2014, Lortholary, 2011). Modern antifungals (AF) improved survival of IPA but lead to ecological, toxic and cost issues. In agreement with the " plan national de la bonne maîtrise des anti-infectieux ", optimization of AF duration in IPA appears therefore challenging.

Positron emission tomography using 2-deoxy-2-[fluorine-18] fluoro- D-glucose integrated with computed tomography (18F-FDG PET/CT) was reported to allow shortened AF duration (Hot, 2011, Chamilos, 2008) and is currently evaluated during chronic disseminated candidiasis {CANHPARI trial, PHRC 2012, NCT01916057}. The investigators raise the hypothesis that normalization of the functional imaging 18F-FDG-PET/CT during IPA could occur earlier than that of conventional imaging. However, due to the current lack of data, an intervention trial evaluating an early AF withdrawal based on 18F-FDG-PET/CT appears premature. In order to optimize IPA treatment duration, a two-step evaluation project has been designed. The first step consists in OPTIFIL prospective project. It will evaluate the therapeutic response through a systematic 18F-FDG-PET/CT at week 6 (crucial time point (Segal) used in recent IPA trials (Marr, 2015, Maertens, 2016). The latter response will be correlated with the kinetics of selected biomarkers including antigens (galactomannan, β-D glucans), circulating Aspergillus DNA and anti-Aspergillus host response markers in addition to the conventional imaging tools obtained at weeks 6 and 12. OPTIFIL project results will serve establishing a decision algorithm used during the second step intervention trial evaluating the accuracy of IPA AF interruption.

Pilot prospective multicenter study of therapeutic follow-up of IPA in patients with hematological malignancy.

Patients will have an inclusion visit (D0) and 8 or 9 follow up visits: D3, W1, W2, W4, W6, End of Treatment, W24 and W48.

Each visit will include physical examination.

Lung CT scan, 18F-FDG-PET/CT, samplings of blood will be performed at different visits in respective centers

β-D-Glucan, Aspergillus fumigatus and Aspergillus spp. quantitative PCRs and host biomarkers such as Aspergillus Elispot will be performed and centralized

Response evaluation will be assessed by an independent committee.

CT response will be evaluated by a blinded radiologist. PET/CT response will be evaluated by 2 blinded nuclear medicine physicians.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years-old
* Patient with hematological malignancy
* Proven or probable invasive pulmonary aspergillosis according to EORTC/MSG modified criteria
* Inclusion ≤ 4 days (≤ 5 days in case of week end) after IPA diagnosis
* Possibility to perform 18F-FDG-PET/CT scanner within the 7 subsequent days following diagnosis
* Informed consent form signed
* Affiliation to French social insurance

Exclusion Criteria:

* Pregnancy or breastfeeding women
* Life expectancy < 3 months
* Fungal or mycobacterial lung co infection at time of IPA diagnosis
* Haematological malignancy with lung location
* Proven or probable mold infection in 6 previous months
* Disseminated aspergillosis (lung and sinus aspergillosis can be included)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Response rate according to 18F-FDG-PET/CT (PET/CT response) | 6 weeks

SECONDARY OUTCOMES:
Response rate according to EORTC/MSG criteria (Segal response). | 6 weeks
Response rate according to EORTC/MSG criteria (Segal response). | 12 weeks
Response rate according to PET/CT | 12 weeks or at the end of treatment
Number of patients for whom 18F-FDG-PET/CT has evidenced extra pulmonary attributable lesions | 6 weeks
Number of patients for whom 18F-FDG-PET/CT has evidenced extra pulmonary attributable lesions | 12 weeks
Number of patients for whom 18F-FDG-PET/CT has evidenced extra pulmonary attributable lesions in initial work-up | first day
Patient mortality rate | 6 weeks
  overall mortality and relationship with Invasive Pulmonary Aspergillosis or Haematological Malignancies
Patient mortality rate | 12 weeks
  overall mortality and relationship with Invasive Pulmonary Aspergillosis or Haematological Malignancies
Patient mortality rate | 24 weeks
  overall mortality and relationship with Invasive Pulmonary Aspergillosis or Haematological Malignancies
Patient mortality rate | 48 weeks
  overall mortality and relationship with Invasive Pulmonary Aspergillosis or Haematological Malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Fanny LANTERNIER, Md, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Olivier LORTHOLARY, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Department of Infectious Diseases and Tropical Medicine, Necker enfants malades hospital, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lortholary O, Gangneux JP, Sitbon K, Lebeau B, de Monbrison F, Le Strat Y, Coignard B, Dromer F, Bretagne S; French Mycosis Study Group. Epidemiological trends in invasive aspergillosis in France: the SAIF network (2005-2007). Clin Microbiol Infect. 2011 Dec;17(12):1882-9. doi: 10.1111/j.1469-0691.2011.03548.x. Epub 2011 Jun 10. PMID 21668573
- [Background] Bitar D, Lortholary O, Le Strat Y, Nicolau J, Coignard B, Tattevin P, Che D, Dromer F. Population-based analysis of invasive fungal infections, France, 2001-2010. Emerg Infect Dis. 2014 Jul;20(7):1149-55. doi: 10.3201/eid2007.140087. PMID 24960557
- [Background] Herbrecht R, Caillot D, Cordonnier C, Auvrignon A, Thiebaut A, Brethon B, Michallet M, Mahlaoui N, Bertrand Y, Preziosi P, Ruiz F, Gorin NC, Gangneux JP. Indications and outcomes of antifungal therapy in French patients with haematological conditions or recipients of haematopoietic stem cell transplantation. J Antimicrob Chemother. 2012 Nov;67(11):2731-8. doi: 10.1093/jac/dks266. Epub 2012 Jul 31. PMID 22850692
- [Background] Baxter CG, Marshall A, Roberts M, Felton TW, Denning DW. Peripheral neuropathy in patients on long-term triazole antifungal therapy. J Antimicrob Chemother. 2011 Sep;66(9):2136-9. doi: 10.1093/jac/dkr233. Epub 2011 Jun 17. PMID 21685202
- [Background] Epaulard O, Villier C, Ravaud P, Chosidow O, Blanche S, Mamzer-Bruneel MF, Thiebaut A, Leccia MT, Lortholary O. A multistep voriconazole-related phototoxic pathway may lead to skin carcinoma: results from a French nationwide study. Clin Infect Dis. 2013 Dec;57(12):e182-8. doi: 10.1093/cid/cit600. Epub 2013 Sep 17. PMID 24046296
- [Background] Tedja R, El-Sherief A, Olbrych T, Gordon S. Multifocal periostitis as a complication of chronic use of voriconazole in a lung transplant recipient. Transpl Infect Dis. 2013 Aug;15(4):424-9. doi: 10.1111/tid.12088. Epub 2013 May 13. PMID 23663268
- [Background] Moon WJ, Scheller EL, Suneja A, Livermore JA, Malani AN, Moudgal V, Kerr LE, Ferguson E, Vandenberg DM. Plasma fluoride level as a predictor of voriconazole-induced periostitis in patients with skeletal pain. Clin Infect Dis. 2014 Nov 1;59(9):1237-45. doi: 10.1093/cid/ciu513. Epub 2014 Jul 3. PMID 24992954
- [Background] Hot A, Maunoury C, Poiree S, Lanternier F, Viard JP, Loulergue P, Coignard H, Bougnoux ME, Suarez F, Rubio MT, Mahlaoui N, Dupont B, Lecuit M, Faraggi M, Lortholary O. Diagnostic contribution of positron emission tomography with [18F]fluorodeoxyglucose for invasive fungal infections. Clin Microbiol Infect. 2011 Mar;17(3):409-17. doi: 10.1111/j.1469-0691.2010.03301.x. PMID 20636432
- [Background] Chamilos G, Macapinlac HA, Kontoyiannis DP. The use of 18F-fluorodeoxyglucose positron emission tomography for the diagnosis and management of invasive mould infections. Med Mycol. 2008 Feb;46(1):23-9. doi: 10.1080/13693780701639546. PMID 18297544
- [Background] Marr KA, Schlamm HT, Herbrecht R, Rottinghaus ST, Bow EJ, Cornely OA, Heinz WJ, Jagannatha S, Koh LP, Kontoyiannis DP, Lee DG, Nucci M, Pappas PG, Slavin MA, Queiroz-Telles F, Selleslag D, Walsh TJ, Wingard JR, Maertens JA. Combination antifungal therapy for invasive aspergillosis: a randomized trial. Ann Intern Med. 2015 Jan 20;162(2):81-9. doi: 10.7326/M13-2508. PMID 25599346
- [Background] Segal BH, Herbrecht R, Stevens DA, Ostrosky-Zeichner L, Sobel J, Viscoli C, Walsh TJ, Maertens J, Patterson TF, Perfect JR, Dupont B, Wingard JR, Calandra T, Kauffman CA, Graybill JR, Baden LR, Pappas PG, Bennett JE, Kontoyiannis DP, Cordonnier C, Viviani MA, Bille J, Almyroudis NG, Wheat LJ, Graninger W, Bow EJ, Holland SM, Kullberg BJ, Dismukes WE, De Pauw BE. Defining responses to therapy and study outcomes in clinical trials of invasive fungal diseases: Mycoses Study Group and European Organization for Research and Treatment of Cancer consensus criteria. Clin Infect Dis. 2008 Sep 1;47(5):674-83. doi: 10.1086/590566. PMID 18637757